CLINICAL TRIAL: NCT07007377
Title: Can the Ergometric Test in Flu-like Syndrome Help in the Outcome Analysis of Unvaccinated Patients
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Pedro Gabriel Senger Braga, PhD, Post-doctoral student, Manager of research from Clinica Pró-Coração, University of Sao Paulo
Other Study IDs: Clínica Pró-Coração
Record Dates: First submitted 2025-03-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Flu-like Syndrome; FLU; Flu-like Symptoms; Vaccination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vaccinated: Vaccinated subjects
  Interventions: Other: Follow-up
- Non-vaccinated: Non-vaccinated subjects
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — Follow-up

SUMMARY:
During the flu-like syndrome, the cardiovascular risk is increased, especially in the elderly. Understanding whether blood pressure assessment during an exercise test can aid in the understanding of patient outcomes, thereby improving prognostic ability in clinical practice, is the focus of the present study. Therefore, the aim of this study is to evaluate the hemodynamic response of adults with flu-like symptoms, both vaccinated and unvaccinated, and to conduct a 30-day follow-up for assessment. Patients who are indicated for an ergometric test and present with flu-like syndrome will be selected. We will inquire about their vaccination history and perform the ergometric test to evaluate test duration, arrhythmias, and ischemias

ELIGIBILITY:
Inclusion Criteria:

* flu-symptoms

Exclusion Criteria:

* recent orthopedic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with flu symptoms, which were vaccinated or not.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Can the ergometric test in flu-like syndrome help in the outcome analysis of unvaccinated patients? | 1 month
  The investigators will analyze whether different responses to exertion, such as blood pressure disorders, are more evident in individuals with or without symptoms who have or have not been vaccinated.

SECONDARY OUTCOMES:
Symptoms | 7 and 14 days after treadmill exercise test
  The investigators will document whether the symptoms are present or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Pró-Coração, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Data protection